CLINICAL TRIAL: NCT05735041
Title: The Efficacy of Computerized Cognitive Training in Patients With Coronary Heart Disease and Cognitive Impairment, no Dementia: a Randomized Controlled Trial
Brief Title: Computerized Cognitive Training in Patients With Coronary Heart Disease and Mild Cognitive Impairment
Acronym: COG-T CHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Beijing Wispirit Technology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Yong Zeng, Professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022BFAZ02
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment; Coronary Heart Disease
Keywords: Cognitive training; Digital therapy
MeSH Terms: conditions — Cognitive Dysfunction; Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive digital therapy group (Experimental): Computer-based cognitive training for 30 minutes at least 5 times a week for 12 weeks; At the end of the 12 weeks, the subjects were randomly divided into two groups. One group continued the training for 12 weeks, at least five times a week for 30 minutes each time, and the other group stopped the training.
  Interventions: Behavioral: Multi-domain cognitive digital therapy
- Positive control group (Active Comparator): Computer-based cognitive training tasks with low or no difficulty variation for 30 minutes at least five times a week for 12 weeks
  Interventions: Behavioral: Basic cognitive therapy

INTERVENTIONS:
Behavioral: Multi-domain cognitive digital therapy — Patients in the cognitive digital therapy group received multi-dimensional targeted cognitive function training electronically, involving attention, memory, executive function, thinking, processing speed and perception. The system will adjust the training difficulty and training plan adaptively according to the patient's current training time and performance, and train the patient's weak cognitive ability as far as possible. The patients had the same total amount of training each day.
  Arms: Cognitive digital therapy group
Behavioral: Basic cognitive therapy — The training content of the positive control group was cognitive training tasks with weak difficulty or no difficulty change. The patients underwent cognitive function training with fixed programs, including 15 training items, and the internal difficulty of the training items remained constant without change. The system presents the training content randomly according to the training scheme. The patients had the same total amount of training each day.
  Arms: Positive control group

SUMMARY:
In this study, a multicentre, double-blind, randomized controlled study based on cognitive training was conducted in patients with coronary heart disease and cognitive impairment but without dementia， to evaluate the effectiveness of computer-based digital therapy in improving the cognitive function of such patients.

DETAILED DESCRIPTION:
This study is a multicentre, double-blind, parallel randomized controlled study using a 1:1 parallel control design. A total of 200 patients with coronary heart disease combined with cognitive decline but no dementia were enrolled in 8 centres. These patients will be randomized to two arms under masking. The intervention arm will receive multi-domain adaptive cognitive training using a tablet. The control arm will receive an active control treatment and use the same tablet to receive the cognitive training tasks with weak difficulty change. Both arms will receive the same intervention dosage for 12 weeks, 5 times a week, and 30 minutes per time. After the 12-week intervention, the intervention arm will be re-randomized into two groups. One group will stop their intervention at 12 weeks; the other group will continue to receive the multi-domain adaptive cognitive training till the 24-week follow-up assessment. The neuro-psychological assessment will be administered at baseline, 12-week, and 24-week assessments for all participants. The structural and functional MRI will be administered at baseline, 12 weeks, and 24 weeks to evaluate the effect of cognitive training on brain structure and function.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 50;
2. Completion of more than 6 years of education;
3. Patients with coronary artery disease confirmed by coronary CT angiography or coronary angiography;
4. Chief complaint of cognitive decline within 1 year;
5. The average score of any cognitive domain in processing speed, situational memory, working memory and visual space measured by the Basic Cognitive Ability Test (BCAT) is less than 1 SD compared with the normal population;
6. Agree to be randomized to cognitive function tests and cognitive training and be able to receive follow-up as required.

Exclusion Criteria:

1. Previous definite diagnosis of dementia or brief Mental State Examination Scale (MMSE) < 24 points;
2. Cognitive dysfunction caused by cranial trauma, cranial tumor, Parkinson's disease, schizophrenia, Alzheimer's disease, anxiety and depression, and other neuropsychiatric diseases;
3. Deaf and mute or other reasons cannot communicate normally;
4. Binge drinking or taking drugs (antihistamines, antipsychotics) that affect cognitive function;
5. Unable to master the use of cognitive training equipment after two 1-hour training instructions each time;
6. Patients who plan to undergo coronary intervention within 6 months or have undergone coronary intervention within 1 month;
7. Severe liver and kidney function injury or critical condition, poor prognosis, estimated survival of less than 1 month.
8. Patients who had received general anesthesia within 3 months;
9. History of stroke and craniocerebral trauma within 6 months;
10. History of Parkinson's disease, schizophrenia, and epilepsy;
11. Prior neurosurgery or history of cranial tumors;
12. Nuclear magnetic examination contraindications: such as metal implants, claustrophobia, etc.;
13. patients living alone;
14. Patients with atrial fibrillation, structural heart disease, and infective endocarditis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Global cognitive function change measured by BCAT in 12 weeks | 12 weeks after randomization
  The proportion of patients whose global cognitive function improves 0.67SD compared to the baseline cognitive function measured by Basic Cognitive Ability test (BCAT). BCAT is a set of neuropsychological battery tests which was designed to measure global cognitive fucntion and cognitive function of sub-domains. Higher scores of BCAT means a better global cognitive function.

SECONDARY OUTCOMES:
Global cognitive function change measured by BCAT in 24 weeks | 24 weeks after randomization
  The proportion of patients whose global cognitive function improves 0.67SD compared to the baseline cognitive function at 24 weeks measured by Basic cognitive Ability Test(BCAT).
Sub-domain cognitive function improvement including memory, attention, and execution memory | 12 weeks, 24 weeks after randomization
  The proportion of patients whose sub-domain cognitive function, including attention, memory, execution function improves measured by the individual capability test in BCAT.
Cognitive score change | 12 weeks, 24 weeks after randomization
  Mean change from baseline in global cognitive function score measured by basic cognitive ability test (BCAT) at 12 weeks and 24 weeks.
Self-efficacy score | 12 weeks, 24 weeks after randomization
  Mean change from baseline in self-efficacy score measured by the General Self-Efficacy Scale at 12 weeks, and 24 weeks
Quality of life score | 12 weeks, 24 weeks after randomization
  Mean change from baseline in the patient's quality of life score measured by EQ-5D-3L at 12 weeks and 24 weeks.
Anxiety score | 12 weeks, 24 weeks after randomization
  Mean change from baseline in the patient's anxiety score at 12 weeks and 24 weeks. Anxiety status will be measured by GAD-7 questionnaire. Higher score of GAD-7 scale represents more anxiety status.
Depression score | 12 weeks, 24 weeks after randomization
  Mean change from baseline in the patient's depression score at 12 weeks and 24 weeks. Depression status will be measured by PHQ-9 questionnaire. Higher score of PHQ-9 scale represents more depression status.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Beijing Anzhen Hospital, Beijing
  - Beijing Sixth Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The second hospital of Chifeng, Chifeng
  - Handan Central Hospital, Handan
  - Inner Mongolia Ordos Central Hospital Kangbashi Department, Ordos
  - The First Affiliated Hospital of Hebei North University, Shijiazhuang
  - The First Hospital of Hebei Medical University, Zhangjiakou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ye Y, Chen Q, Li R, Wang X, Sun Y, Li F, Liu X, Wang L, Ning X, Tian H, Zhao W, Ma C, Zhang H, Zeng Y. The efficacy of computerized cognitive training in patients with coronary heart disease and cognitive impairment, no dementia: study protocol for a randomized controlled trial. Trials. 2025 Feb 21;26(1):64. doi: 10.1186/s13063-025-08745-6. PMID 39985041

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-01-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT05735041/SAP_000.pdf